CLINICAL TRIAL: NCT05692531
Title: Optimizing Study Design to Test a Community-level Intervention to Reduce Intersectional Stigma and Increase HIV Testing and Prevention Among African-American/Black MSM
Brief Title: Evaluation of A Story Within A Story: The Novel CHHARGE Intervention Component
Acronym: CHHARGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: City University of New York (Other)
Responsible Party: Principal Investigator, Victoria Frye, Medical Professor, City University of New York
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R34MH121295 (NIH)
Record Dates: First submitted 2022-12-22; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Intersectional Stigma

STUDY DESIGN:
Intervention Model Description: This is an evaluation of a virtual event. The investigators will conduct a social media metrics analysis (of the social media-based run-up to the event as well as the actual event) via responses to polls embedded within the social media-based run-up, and sentiment assessment and analysis during the event itself. The investigators will conduct "flash polls" during the event using sentiments that reflect key stigmatization process-related aspects of the scenarios being depicted, for example asking attendees to rate the actors on specific qualities on a scale of 1 to 10 (for example, "respect" "admire" "dislike" "annoyed" "tactful" "sensitive" "shady" etc.); the investigators will repeat this after the scenarios are screened and integrate the immediate results into the discussion of the filmed scenarios. The investigators will conduct flash polls on confidence confronting stigmatizing language toward someone who is considering taking PrEP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Story Within A Story (Experimental): This is a single event that will be evaluated using quasi-experimental design methods.
  Interventions: Behavioral: A Story Within A Story

INTERVENTIONS:
Behavioral: A Story Within A Story — The intervention is the screening via Zoom of "A Story Within A Story," two dramatized scenarios. The first depicts a reinforcing feedback loop connecting internalized, anticipated and enacted HIV stigma and serosorting within the Black SGL/MSM community. Set during the COVID-19 pandemic, it depicts a Zoom call among three generations of Black SGL/MSM, a chosen family. In this scene, the oldest member of the family, not knowing that the youngest has just tested positive for HIV, describes how they would never partner with someone who was living with HIV because of what they saw at the beginning of the HIV epidemic. The middle-aged member attempts to mitigate the damage done by this, while the youngest member describes what kind of support he needs. The second scenario depicts a Telehealth visit between a young Black gay man and his sexual health provider; his older lover joins the call at one point and the focus is on sexual communication and PrEP use.
  Other Names: CHHARGE novel component

SUMMARY:
Using a quasi-experimental evaluation approach, the purpose of this study is to assess feasibility, acceptability, and preliminary efficacy of a novel community-level intervention component, which is a filmed dramatization or set of "scenarios" to be "screened" in a virtual event. Attendees will be polled and engaged in an evaluation of the scenarios, before during and after the screening. This NCT registration is for the final aim of the study as described in the detailed description (AIMS) below. (Please note Aims 1-2 are complete.)

DETAILED DESCRIPTION:
Increasing access to and uptake of consistent HIV testing and biomedical prevention is critical to ending the epidemic in the United States (US) among gay, bisexual and other men who have sex with other men (MSM). This is particularly true for urban, African-American/Black MSM, who are disproportionately affected by HIV/AIDS in the US2-4 and would thus benefit from consistent testing, which is the gateway to treatment and prevention. NYC is the metropolitan area in the US with the largest number of newly diagnosed HIV infections among MSM and 89-94% of all people living with HIV/AIDS (PLWHA) in the US reside in urban areas. HIV stigma is a key barrier to HIV treatment and prevention, reducing access to testing and anti-retroviral treatment (ART). Stigmas specific to biomedical prevention (e.g., PrEP/PEP stigma) and HIV testing have emerged and influence intentions to use PrEP/PEP and testing. In addition, homophobia has been identified as a barrier to prevention access, with structural homophobia negatively associated with PEP awareness and PrEP use. Intersectional HIV-related stigmas and homophobia may be especially significant barriers to HIV testing and prevention among African-American/Black MSM, who test less often and are more likely to live with undiagnosed HIV/AIDS compared with white MSM. African-American/Black MSM live in a racist society, which operates at the personal and institutional levels. This results in experiences of HIV-related stigma and homophobia being racialized, further inhibiting access to and uptake of testing, prevention and treatment.

Interventions to decrease HIV stigma have aimed primarily at the individual level and on internalized stigma and/or personal attitudes, providing education and increased contact with PLWHA to reduce stereotyping and active discrimination. Few have addressed HIV stigma and homophobia simultaneously or at the community level. One exception, designed and evaluated by study team leaders, Frye & Taylor-Akutagawa, is CHHANGE (Challenge HIV/AIDS Stigma & Homophobia and Gain Empowerment; R21 MH102182-01; PI: Frye), a community-level, theory-based, anti-stigma and -homophobia intervention. Designed for African-American urban neighborhoods with high HIV prevalence, and broadly framed within socioecological, empowerment and stigma theories, CHHANGE focused on: enhancing visibility; increasing contact with LGBTQ people and PLWHA; educating on stigmatization processes and effects; enhancing empathy and perspective-taking; challenging stereotyped beliefs; raising critical consciousness; and teaching skills to analyze and interrupt stigma & homophobia in organizations, families and individuals. Results of the quasi-experimental, matched-community study found that HIV testing increased by 350% at the intervention community site, though changes in community-level HIV stigma and homophobia were not statistically significant across communities.

The emergence of PEP/PrEP and testing stigmas highlight a gap in our HIV testing and prevention toolbox for MSM of color and a need for interventions that address intersectional stigmas. To our knowledge, no intervention addresses intersectional HIV, PrEP/PEP, testing stigmas, and homophobia, in the context of racism. To address this gap, the investigators propose an R34 to adapt and enhance CHHANGE to simultaneously address intersectional stigmas and plan a trial to test the community-level intervention.

The Specific Aims are:

1. Inform design of novel components specific to PrEP/PEP and testing stigma. The investigators will conduct group model building (GMB), a systems science technique, with community residents and African-American/Black MSM (N=80) to understand the intersectional complexity of HIV-related stigmas, homophobia, and racism, in context, and identify novel levers that may influence consistent HIV testing and prevention uptake.
2. Systematically adapt the CHHANGE intervention to integrate novel anti-stigma, -homophobia, and -racism content and activities (re-named CHHARGE: Challenge HIV Stigma, Homophobia and Racism and Gain Empowerment) and plan a pilot using optimal study design methods. The investigators will ideate, prototype and component test (N=30), using design thinking and traditional adaptation methods, novel modules and components in the community. With input from a Senior Advisory Board (SAB), the investigators will identify optimal study design features (around areal boundaries, "big data" outcome measures, sampling, contamination, lagged effects) for planning a trial of the community-level intervention (e.g., a community cluster randomized trial).
3. Assess feasibility, acceptability, and preliminary efficacy of novel component. The investigators will conduct a quasi-experimental evaluation to assess feasibility of the novel component. The investigators will assess preliminary efficacy of the component in reducing community-level stigmas (HIV, PrEP/PEP, testing) by increasing likelihood of engaging in stigma interrupting communication and behavior, particularly as related to the theoretical targets identified via Phases 1 and 2, as well as likelihood of consistent HIV testing and PrEP/PEP uptake.

Thus far, the research has completed phases 1 and 2 in partnership with Mobilizing Our Brother Initiative (MOBI) creating an innovative module that facilitates consistent HIV testing, and access to, uptake of and adherence to new biomedical HIV prevention modalities, with the goal of lowering community-level viral load and ultimately a diminution of the HIV epidemic among urban, Black MSM in the US.

ELIGIBILITY:
Inclusion Criteria:

* all attendees of the event

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
internalized/anticipated HIV stigma | immediately post-intervention
  single-item, adapted, self-reported internalized/anticipated HIV stigma; we will use an item from Sayles et al (2008) valid and reliable measure of internalized/anticipated stigma (for example "I am living with HIV and feel ashamed when I tell people that I have HIV/I am not living with HIV but would feel ashamed if I had to tell people that I have HIV"). This item is adapted from Sayles, J. N., Hays, R. D., Sarkisian, C. A., Mahajan, A. P., Spritzer, K. L., & Cunningham, W. E. (2008). Development and psychometric assessment of a multidimensional measure of internalized HIV stigma in a sample of HIV-positive adults. AIDS and Behavior, 12(5), 748-758.
internalized homophobia | immediately post-intervention
  single-item, self-reported internalized HIV stigma; we will use items from a valid and reliable measure of internalized homophobia (Smolenski et al 2010; for example "I would change myself to be heterosexual, if I could") From: Smolenski, D. J., Diamond, P. M., Ross, M. W., & Rosser, B. S. (2010). Revision, criterion validity, and multigroup assessment of the Reactions to Homosexuality Scale. Journal of Personality Assessment,92, 568-576
internalized/anticipated PrEP stigma | immediately post-intervention
  single-item, self-reported PrEP stigma; we will use an item from a measure of PrEP stigma (Frye et al 2020) (for example "People who who use PrEP are having too much sex or sex with the wrong kinds of people") From: Chittamuru, D., Frye, V., Koblin, B. A., Brawner, B., Tieu, H. V., Davis, A., & Teitelman, A. M. (2020). PrEP stigma, HIV stigma, and intention to use PrEP among women in New York City and Philadelphia. Stigma and health, 5(2), 240.
HIV testing stigma | immediately post-intervention
  single-item, self-reported HIV testing stigma; we will use an item adapted from a measure of HIV testing stigma (for example "if people know I get HIV tests frequently, they will think I am promiscuous or am having sex with men") From: Andrinopoulos, K., Hembling, J., Guardado, M. E., de Maria Hernández, F., Nieto, A. I., & Melendez, G. (2015). Evidence of the negative effect of sexual minority stigma on HIV testing among MSM and transgender women in San Salvador, El Salvador. AIDS and Behavior, 19(1), 60-71.

IPD SHARING:
Plan to Share IPD: Undecided
Because this is a quasi-experimental evaluation of an event, it is unclear if the data would be of any use to any other researchers other than this team.